CLINICAL TRIAL: NCT01240772
Title: Cost-effectiveness of New Surgical Treatments for Haemorrhoidal Disease - Randomized Controlled Trial Comparing Transanal Doppler-guided Arterial Ligation With Mucopexy and Stapled Haemorrhoidopexy (Longo's Technique)
Brief Title: Randomized Controlled Trial Comparing Transanal Doppler-guided Arterial Ligation With Mucopexy and Stapled Haemorrhoidopexy
Acronym: LIGALONGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STIC/10/01; IDRCB 2010-A00642-37 (Other: Afssaps)
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Symptomatic Haemorrhoidal Disease Requiring Surgical Management
Keywords: Haemorrhoids, Surgery, Cost-effectiveness, Morbidity, Risk assessment,RCT, Stapled haemorrhoidopexy, Doppler-guided, Haemorrhoidal artery ligation, Outcome
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DGALM (Experimental): doppler-guided arterial ligation with mucopexy
  Interventions: Device: doppler-guided arterial ligation with mucopexy
- SH (Active Comparator): stapled haemorrhoidopexy according to Longo
  Interventions: Device: stapled haemorrhoidopexy according to Longo

INTERVENTIONS:
Device: doppler-guided arterial ligation with mucopexy — doppler-guided arterial ligation with mucopexy
  Other Names: THD; AMI
  Arms: DGALM
Device: stapled haemorrhoidopexy according to Longo — stapled haemorrhoidopexy according to Longo
  Arms: SH

SUMMARY:
This multicentre RCT aims to compare two surgical treatments of haemorrhoidal disease: doppler-guided arterial ligation with mucopexy (DGALM) and stapled haemorrhoidopexy according to Longo (SH). The hypothesis of the trial is that the DGALM is at a lesser risk and is more cost-effective than SH. With a large number of patients managed in more than 20 centres, we aim to demonstrate that DGALM has a lower morbidity than SH when treating haemorrhoidal disease. At a lower postoperative risk and a lower risk of sequelae, the DGALM would demonstrate to be cost-effective for health care system and attractive for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) 18 - 75 y.o
* Suffering from symptomatic grade II or III haemorrhoidal disease (bleeding and/or prolapse)
* requiring surgery

Exclusion Criteria:

* Acute complication of haemorrhoidal disease
* History of anal surgery for haemorrhoids
* Congenital or acquirred anal stenosis
* Anal fissure or perianal abcess
* Inflammatory bowel disease
* Colon or rectal cancerv History of rectal or sigmoid resection
* Rectal prolapse
* Portal vein hypertension
* Haemophylia
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Morbidity at 60 days postoperatively of the 2 techniques | 60-90 days
  Morbidity at 60 days postoperatively of the 2 techniques, the morbidity being defined as " the sum of adverse events that occurred during or after the procedure for a period of 2 months".Primary outcome measure is "the percentage of patients with complication, whatever the number of complications per patient and the grade of complication according to the Clavien-Dindo classification".

SECONDARY OUTCOMES:
Cost-effectiveness of the 2 procedures | 12 months
  global cost of the treatment, length of stay, sick leave, cost of complications and sequelae management
Success rate at 1 year of each procedure regarding the control of haemorrhoids symptoms | 1 year
  Efficiency regarding the cure of haemorrhoidal symptoms that led to surgery
  * Pain
  * Persisting or recurring symptoms of haemorrhoidal disease
  * Prolapse
  * Bleeding
  * Haemorrhoidal thrombose
  * Occurrence of new anal symptoms / surgical sequelae
  * Incontinence
  * Soiling
  * Pruritus
  * Anal stenosis
  * Constipation
  * Fissure
  * Other rare complication
Rate of anatomical or functional sequelae | 1 year
  Assessment will be done according to Grade II vs Grade III patients as well as patients without and with antithrombotic treatments

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - Angers University Hospital, Angers
  - Grenoble University Hospital, Grenoble
  - La Roche/Yon Hospital, La Roche/Yon
  - Lille University Hospital "Claude Huriez", Lille
  - Marseille University Hospital "Hôpital Nord", Marseille
  - Marseille University Hospital "La Timone", Marseille
  - Nantes University Hospital, Nantes
  - Niort Hospital, Niort
  - Nîmes University Hospital, Nîmes
  - Polyclinic H. MALARTIC, Ollioules
  - "Institut Mutualiste Montsouris", Paris
  - Hopital St Joseph, Paris
  - Poissy / Saint-Germain en Laye Hospital, Poissy
  - Rennes University Hospital, Rennes
  - Saint-Etienne University Hospital, Saint-Etienne
  - "Pôle Hospitalier Mutualiste", Saint-Nazaire
  - Strasbourg University Hospital, Strasbourg
  - Foch Hospital, Suresnes
  - Talence Bagatelle Hospital, Talence
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours
  - Vichy Hospital, Vichy

REFERENCES:
- [Derived] Woaye-Hune P, Hardouin JB, Lehur PA, Meurette G, Vanier A. Practical issues encountered while determining Minimal Clinically Important Difference in Patient-Reported Outcomes. Health Qual Life Outcomes. 2020 May 27;18(1):156. doi: 10.1186/s12955-020-01398-w. PMID 32460882
- [Derived] Venara A, Podevin J, Godeberge P, Redon Y, Barussaud ML, Sielezneff I, Queralto M, Bourbao C, Chiffoleau A, Lehur PA; LigaLongo Study Group. A comparison of surgical devices for grade II and III hemorrhoidal disease. Results from the LigaLongo Trial comparing transanal Doppler-guided hemorrhoidal artery ligation with mucopexy and circular stapled hemorrhoidopexy. Int J Colorectal Dis. 2018 Oct;33(10):1479-1483. doi: 10.1007/s00384-018-3093-8. Epub 2018 May 28. PMID 29808305